CLINICAL TRIAL: NCT01933594
Title: A Phase I/II Study of Romidepsin in HIV-Infected Adults With Suppressed Viremia on Antiretroviral Therapy to Assess Safety, Tolerability, and Activation of HIV-1 Expression
Brief Title: Evaluating the Safety and Efficacy of Romidepsin in Combination With Antiretroviral Therapy in HIV-Infected Adults With Suppressed Viral Load
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5315; 11892 (Registry Identifier: DAIDS-ES); ACTG 5315
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — romidepsin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1-Arm 1A (Romidepsin) (Experimental): Participants in Cohort 1, Arm 1A received Romidepsin intravenously (IV) over 4 hours (beginning at Hour 0) at the Day 0 study visit. Dose of Romidepsin was 0.5 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Romidepsin
- Cohort 1-Arm 1B (Placebo for Romidepsin) (Placebo Comparator): Participants in Cohort 1, Arm 1B received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0 study visit. Dose of sodium chloride for injection placebo was 0.5 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Placebo for Romidepsin
- Cohort 2-Arm 2A (Romidepsin) (Experimental): Participants in Cohort 2, Arm 2A received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0 study visit. Dose of Romidepsin was 2 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Romidepsin
- Cohort 2-Arm 2B (Placebo for Romidepsin) (Placebo Comparator): Participants in Cohort 2, Arm 2B received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0 study visit. Dose of sodium chloride for injection placebo was 2 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Placebo for Romidepsin
- Cohort 3-Arm 3A (Romidepsin) (Experimental): Participants in Cohort 3, Arm 3A received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0 study visit. Dose of Romidepsin was 5 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Romidepsin
- Cohort 3-Arm 3B (Placebo for Romidepsin) (Placebo Comparator): Participants in Cohort 3, Arm 3B received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0 study visit. Dose of sodium chloride for injection placebo was 5 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Placebo for Romidepsin
- Cohort 4-Arm 4A (Romidepsin) (Experimental): Participants in Cohort 4, Arm 4A received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0, 14, 28, and 42 study visits. Dose of Romidepsin was 5 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Romidepsin
- Cohort 4-Arm 4B (Placebo for Romidepsin) (Placebo Comparator): Participants in Cohort 4, Arm 4B received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0, 14, 28, and 42 study visits. Dose of sodium chloride for injection placebo was 5 mg/m^2, with total dose based on the participant's body surface area (determined by participant's height and weight).
  Interventions: Drug: Placebo for Romidepsin

INTERVENTIONS:
Drug: Romidepsin — RMD administered over 4 hours via an intravenous (IV) catheter.
  Other Names: RMD; Istodax
  Arms: Cohort 1-Arm 1A (Romidepsin); Cohort 2-Arm 2A (Romidepsin); Cohort 3-Arm 3A (Romidepsin); Cohort 4-Arm 4A (Romidepsin)
Drug: Placebo for Romidepsin — Placebo for RMD administered over 4 hours via an IV catheter.
  Other Names: 0.9% NaCl; 0.9% sodium chloride
  Arms: Cohort 1-Arm 1B (Placebo for Romidepsin); Cohort 2-Arm 2B (Placebo for Romidepsin); Cohort 3-Arm 3B (Placebo for Romidepsin); Cohort 4-Arm 4B (Placebo for Romidepsin)

SUMMARY:
Antiretroviral therapy (ART) can reduce HIV to very low levels in the blood, but it cannot cure HIV infection because a small amount of virus remains in cells as a hidden (latent) form. The purpose of this study was to evaluate the safety and efficacy of single dose and multiple dose administration of romidepsin (RMD) in HIV-infected adults.

DETAILED DESCRIPTION:
A major challenge in eradicating HIV-1 infection is the persistence of virus in long-lived cells, such as latently infected memory CD4 T cells. One approach for eliminating the HIV-1 reservoir is to activate viral replication in these latently infected CD4 T cells by targeting cellular mechanisms that repress proviral transcription. Histone deacetylase inhibitors (HDACis), such as RMD, induce HIV-1 expression by increasing acetylation and facilitating transcriptional activation of HIV-1. RMD administered in combination with ART may serve as an important component of a strategy to eradicate the HIV-1 latent reservoir. The purpose of this study was to evaluate the safety and efficacy of single dose and multiple dose administration of RMD in HIV-infected adults.

Participants were sequentially enrolled into four cohorts and randomly assigned to receive either RMD or placebo. The cohorts differed in the dose of RMD given. Participants in Cohorts 1, 2, and 3 had one intravenous (IV) infusion of RMD or placebo at Day 0. Participants in Cohort 4 had four IV infusions of RMD or placebo at Days 0, 14, 28, and 42.

For participants in Cohorts 1, 2, and 3, study duration was 4 weeks. For participants in Cohort 4, study duration was a minimum of 24 weeks and a maximum of 48 weeks.

Participants attended several study visits, which could include a physical examination, blood and urine collection, pharmacokinetic (PK) sampling, and an electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria: Cohorts 1, 2, & 3

* HIV-1 infection, documented by any licensed rapid HIV test or HIV E/CIA test kit at any time prior to study entry & confirmed by a licensed Western blot or a 2nd antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA
* Receiving 2 (or more) nucleoside or nucleotide reverse transcriptase inhibitors with raltegravir, dolutegravir, or efavirenz for at least 90 days prior to study entry with no intention to change for the duration of the study
* Documentation of at least 2 historical HIV-1 RNA measurements <50 copies/mL while on ART obtained by standard ultrasensitive assay. Documentation of the 1st measurement must be from a result obtained between 365-91 days, inclusive, prior to study entry. Documentation of the 2nd measurement must be from a result obtained between 730-366 days, inclusive, prior to study entry. In addition, there must be no HIV-1 RNA values ≥50 copies/mL for at least 365 days prior to study entry.
* CD4 cell count ≥300 cells/mm^3 obtained within 90-50 days prior to study entry at any US laboratory that has a CLIA certification or equivalent
* HIV-1 RNA level of <50 copies/mL obtained by standard ultrasensitive assay within 90-50 days prior to study entry
* HIV-1 RNA level of ≥0.4 copies/mL obtained by SCA within 90-50 days prior to study entry. This result must be available prior to the pre-entry visit
* The following laboratory values obtained within 21-0 days prior to study entry by any laboratory that has a CLIA certification or equivalent

  * ANC ≥1500 cells/mm^3
  * Hemoglobin ≥12.0 g/dL for men & >11.0 g/dL for women
  * Platelet count ≥120,000/mm^3
* The following laboratory values obtained within 21-7 days prior to study entry by any laboratory that has a CLIA certification or equivalent

  * CrCl ≥60 mL/min
  * Potassium & magnesium within normal limits
  * AST (SGOT) <2.0 x ULN
  * ALT (SGPT) <2.0 x ULN
  * Alkaline phosphatase <2.0 x ULN
  * Total bilirubin <2.5 x ULN
* HCV antibody negative result within 90-50 days prior to study entry or, for study candidates who are HCV antibody positive (based on testing performed at any time prior to study entry), a negative HCV RNA result obtained within 90-50 days prior to study entry
* Negative HBsAg result obtained within 90-50 days prior to study entry or a positive HBsAb result at any time prior to study entry
* For females of reproductive potential, negative serum or urine pregnancy test (latter with sensitivity of ≤25 mIU/mL) at the screening visit, pre-entry visit within 21-7 days prior to study entry, & at entry prior to romidepsin infusion, by any US laboratory that has a CLIA certification or equivalent
* Female candidates of reproductive potential must refrain from participating in active attempts to become pregnant, &, if participating in sexual activity that could lead to pregnancy, must agree to use at least 2 reliable forms of contraception that are non-estrogen based. All female participants of reproductive potential must be instructed to use contraceptives for 6 months/180 days after completing RMD or placebo infusion
* Karnofsky performance score ≥80 within 21-7 days prior to study entry
* Men and women age ≥ 18 years
* Ability & willingness to provide written informed consent
* Investigator anticipates that a fully active alternative ART regimen could be constructed in the event of virologic failure on the current ART regimen

Exclusion Criteria: Cohorts 1, 2, & 3

* History of or current malignancy requiring cytotoxic therapy
* Bacterial, fungal, or viral infection (other than HIV) requiring systemic therapy within 30 days prior to entry
* History of or current CMV end organ disease (eg, retinitis)
* History of or current AIDS-related syndromes or symptoms that pose a perceived excessive risk for study drug-related morbidity, as determined by the investigator
* Chronic, acute, or recurrent infections that are current & serious in the opinion of the investigator & for which the participant has not completed at least 14 consecutive days of therapy within 30 days prior to study entry and/or is not clinically stable
* Active autoimmune disorders including but not limited to: inflammatory bowel diseases, scleroderma, severe psoriasis as determined by the investigator, systemic lupus erythematosus, rheumatoid arthritis & optic neuritis
* History of seizure disorders
* History of anticonvulsant use within 60 days prior to study entry
* History of MI within 6 months prior to study entry, history of QTc prolongation (defined as ECG with QTc intervals >450 ms) at any time prior to study entry, NYHA class III or IV heart failure at any time prior to study entry, or family history of prolonged QTc syndrome
* Breastfeeding
* Use of immunomodulators (eg, interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry
* Any vaccination within 30 days prior to entry or intent to receive an elective vaccination (eg, flu shot, hepatitis A or B vaccine) during the course of the study
* Intent to use cytokines (e.g., IL-2 or IL-12) during the course of the study. Prior administration of cytokines is not an exclusion criterion; however, at least 60 days between the most recent cycle of any cytokine and study entry is required
* Within 60 days prior to study entry, use of systemic azole antifungals (voriconazole, itraconazole, ketoconazole); dexamethasone; macrolide antibiotics (azithromycin, clarithromycin, erythromycin); ARVs that are inhibitors of, or are metabolized by, CYP3A4 (atazanavir, ritonavir, nelfinavir, indinavir, saquinavir, darunavir, lopinavir, rilpivirine, maraviroc); cobicistat; warfarin; nefazodone; rifamycins (rifabutin, rifampin, rifapentine); St. John's Wort; carbamazepine; phenytoin; phenobarbital; amiodarone; dofetilide; pimozide; procainamide; quinidine; sotalol; & birth control products containing estrogen; drugs that are p-glycoprotein inhibitors; & drugs that prolong the QTc interval with a risk of Torsades de Pointes
* Known allergy, sensitivity, or any hypersensitivity to components of RMD or its formulation
* Use of histone deacetylase inhibitors (eg, vorinostat, valproic acid) at any time prior to study entry
* Active illicit drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Acute or serious illness requiring systemic treatment and/or hospitalization that is not resolved within 30 days prior to entry
* Psychosocial conditions that would prevent study compliance and follow-up, as determined by the investigator
* Documented opportunistic infections within 60 days prior to entry

Inclusion Criteria: Cohort 4, Step 1

* HIV-1 infection, documented by any licensed rapid HIV test or HIV E/CIA test kit at any time prior to study entry & confirmed by a licensed Western blot or a 2nd antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA
* Receiving 2 or more nucleoside or nucleotide reverse transcriptase inhibitors with raltegravir or dolutegravir for at least 90 days prior to study entry with no intention to change for the duration of the study
* Documentation of at least 2 historical HIV-1 RNA measurements <50 copies/mL while on ART obtained by standard ultrasensitive assay. Documentation of the first measurement must be from a result obtained between 365-61 days, inclusive, prior to study entry. Documentation of the second measurement must be from a result obtained between 730-366 days, inclusive, prior to study entry. In addition, there must be no HIV-1 RNA values ≥50 copies/mL for at least 365 days prior to study entry
* CD4 cell count ≥300 cells/mm^3 obtained between 36-60 days prior to study entry (screening visit) at any US laboratory that has a CLIA certification or equivalent
* HIV-1 RNA level of <50 copies/mL obtained by standard ultrasensitive assay at screening (between 36-60 days prior to study entry)
* The following laboratory values obtained at pre-entry (between 3-14 days prior to study entry) by any laboratory that has a CLIA certification or equivalent

  * ANC ≥1500 cells/mm^3
  * Hemoglobin ≥12.0 g/dL for men & >11.0 g/dL for women
  * Platelet count ≥120,000/mm^3
  * CrCl ≥60 mL/min
  * Potassium & magnesium within normal limits
  * AST (SGOT) <2.0 x ULN
  * ALT (SGPT) <2.0 x ULN
  * Alkaline phosphatase <2.0 x ULN
  * Total bilirubin <2.5 x ULN
* HCV antibody negative result at screening (between 36-60 days prior to study entry) or, for study candidates who are HCV antibody positive (based on testing performed at any time prior to study entry), a negative HCV RNA result obtained at screening
* Negative HBsAg result obtained at screening (between 36-60 days prior to study entry) or a positive HBsAb result at any time prior to study entry
* For females of reproductive potential, negative urine pregnancy test (with a sensitivity of ≤25 mIU/mL) at screening (between 36-60 days prior to study entry), at pre-entry (between 3-14 days prior to study entry), & at entry prior to infusion, by any US laboratory that has a CLIA certification or equivalent
* Female candidates of reproductive potential must refrain from participating in active attempts to become pregnant, &, if participating in sexual activity that could lead to pregnancy, must agree to use at least 2 reliable forms of contraception that are non-estrogen based. All participants of reproductive potential will be instructed to use contraceptives for 6 months or 180 days after completing RMD/placebo infusion
* Karnofsky performance score ≥80 at pre-entry (between 3-14 days prior to study entry)
* Men and women age ≥ 18 years
* Ability & willingness to provide written informed consent
* Investigator anticipates that a fully active alternative ART regimen could be constructed in the event of virologic failure on the current ART regimen

Exclusion Criteria: Cohort 4, Step 1

* History of or current malignancy requiring cytotoxic therapy
* Bacterial, fungal or viral infection (other than HIV) requiring systemic therapy within 30 days prior to entry
* History of or current CMV end organ disease (eg, retinitis)
* History of or current AIDS-related syndromes or symptoms that pose a perceived excessive risk for study drug-related morbidity, as determined by the investigator
* Chronic, acute, or recurrent infections that are current & serious, in the opinion of the investigator, for which the participant has not completed at least 14 consecutive days of therapy within 30 days prior to study entry and/or is not clinically stable
* Active autoimmune disorders including but not limited to inflammatory bowel diseases, scleroderma, severe psoriasis as determined by the investigator, systemic lupus erythematosus, rheumatoid arthritis, & optic neuritis
* History of seizure disorders
* History of anticonvulsant use within 60 days prior to study entry
* History of MI within 6 months prior to study entry, history of QTc prolongation (defined as ECG with QTc intervals >450 ms) at any time prior to study entry, NYHA class III or IV heart failure at any time prior to study entry, or family history of prolonged QTc syndrome
* Breastfeeding
* Use of immunomodulators (eg, interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry
* Any vaccination within 30 days prior to entry or intent to receive an elective vaccination (eg, flu shot, hepatitis A or B vaccine) during the course of the study
* Intent to use cytokines (eg, IL-2 or IL-12) during the course of the study
* Within 60 days prior to study entry, use of systemic azole antifungals (voriconazole, itraconazole, ketoconazole), dexamethasone, macrolide antibiotics (azithromycin, clarithromycin, erythromycin), antiretrovirals that are inhibitors of, or are metabolized by CYP3A4 (atazanavir, ritonavir, nelfinavir, indinavir, saquinavir, darunavir, lopinavir, rilpivirine, maraviroc), cobicistat, warfarin, nefazodone, rifamycins (rifabutin, rifampin, rifapentine), St. John's Wort, carbamazepine, phenytoin, phenobarbital, amiodarone, dofetilide, pimozide, procainamide, quinidine, sotalol, & birth control products containing estrogen, drugs that are p-glycoprotein inhibitors, & drugs that prolong the QTc interval with a risk of Torsades de Pointes
* Known allergy/sensitivity or any hypersensitivity to components of RMD or its formulation
* Use of histone deacetylase inhibitors (eg, vorinostat, valproic acid) at any time prior to study entry
* Active illicit drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Acute or serious illness requiring systemic treatment and/or hospitalization that is not resolved within 30 days prior to entry
* Psychosocial conditions that would prevent study compliance & follow-up as determined by the investigator
* Documented opportunistic infections within 60 days prior to entry
* Use of any of the medications listed in the Prohibited Medications table in the protocol

See the protocol for Inclusion and Exclusion Criteria for Cohort 4, Steps 2, 3, and 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mellors, MD, Study Chair — University of Pittsburgh; Deborah McMahon, MD, Study Chair — University of Pittsburgh
Locations (10):
- United States (10):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Ylisastigui L, Archin NM, Lehrman G, Bosch RJ, Margolis DM. Coaxing HIV-1 from resting CD4 T cells: histone deacetylase inhibition allows latent viral expression. AIDS. 2004 May 21;18(8):1101-8. doi: 10.1097/00002030-200405210-00003. PMID 15166525
- [Background] Klimek VM, Fircanis S, Maslak P, Guernah I, Baum M, Wu N, Panageas K, Wright JJ, Pandolfi PP, Nimer SD. Tolerability, pharmacodynamics, and pharmacokinetics studies of depsipeptide (romidepsin) in patients with acute myelogenous leukemia or advanced myelodysplastic syndromes. Clin Cancer Res. 2008 Feb 1;14(3):826-32. doi: 10.1158/1078-0432.CCR-07-0318. PMID 18245545
- [Derived] McMahon DK, Zheng L, Cyktor JC, Aga E, Macatangay BJ, Godfrey C, Para M, Mitsuyasu RT, Hesselgesser J, Dragavon J, Dobrowolski C, Karn J, Acosta EP, Gandhi RT, Mellors JW. A Phase 1/2 Randomized, Placebo-Controlled Trial of Romidespin in Persons With HIV-1 on Suppressive Antiretroviral Therapy. J Infect Dis. 2021 Aug 16;224(4):648-656. doi: 10.1093/infdis/jiaa777. PMID 34398236
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014. Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1-Arm 1A (Romidepsin): Participants in Cohort 1, Arm 1A received Romidepsin intravenously (IV) over 4 hours (beginning at Hour 0) at the Day 0 study visit.
- Cohort 2-Arm 2A (Romidepsin): Participants in Cohort 2, Arm 2A received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0 study visit.
- Cohort 3-Arm 3A (Romidepsin): Participants in Cohort 3, Arm 3A received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0 study visit.
- Cohorts 1-3 (Placebo for Romidepsin): Participants in Cohorts 1-3, received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0 study visit.
- Cohort 4-Arm 4A (Romidepsin): Participants in Cohort 4, Arm 4A received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0, 14, 28, and 42 study visits.
- Cohort 4-Arm 4B (Placebo for Romidepsin): Participants in Cohort 4, Arm 4B received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0, 14, 28, and 42 study visits.
Period: Overall Study
Arm/Group | Cohort 1-Arm 1A (Romidepsin) | Cohort 2-Arm 2A (Romidepsin) | Cohort 3-Arm 3A (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin) | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Started | 12 | 12 | 12 | 7 | 13 | 3
Completed | 11 | 12 | 12 | 7 | 11 | 3
Not Completed | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Ineligible for subsequent study step | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants. The placebo arms of Cohorts 1-3 were combined for the Baseline Characteristics.
Groups:
- Cohorts 1-3 (Placebo for Romidepsin): Participants in Cohorts 1-3 who received 0.9% sodium chloride for injection IV over 4 hours (beginning at Hour 0) at the Day 0 study visit.
- Total: Total of all reporting groups
Arm/Group | Cohort 1-Arm 1A (Romidepsin) | Cohort 2-Arm 2A (Romidepsin) | Cohort 3-Arm 3A (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin) | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 7 | 13 | 3 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 11 | 6 | 11 | 3 | 55
  >=65 years | 0 | 0 | 1 | 1 | 2 | 0 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [29 to 54] | 52 [44 to 54] | 51 [37 to 58] | 51 [44 to 56] | 56 [48 to 61] | 45 [34 to 53] | 52 [41 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 4 | 1 | 8
  Male | 11 | 11 | 11 | 7 | 9 | 2 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 8 | 8 | 6 | 5 | 6 | 2 | 35
  Black non-Hispanic | 4 | 3 | 5 | 2 | 6 | 1 | 21
  Hispanic (regardless of race) | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian, Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 12 | 7 | 13 | 3 | 59
Baseline SCA in Cohorts 1-3 [Median (Inter-Quartile Range); unit: log10 copies/mL] — Baseline HIV-1 RNA levels as detected by single copy assay (SCA) was calculated as the average of the pre-entry and entry SCA measurements for Cohorts 1-3 Population: Cohorts 1-3 were analyzed separately from Cohort 4
  log10 copies/mL
    number analyzed (Participants) | 12 | 12 | 12 | 7 | 0 | 0 | 43
    (all) | 0.08 [-0.13 to 0.32] | -0.2 [-0.49 to 0.02] | 0.22 [-0.6 to 0.57] | 0.38 [0.22 to 0.51] |  |  | NA [NA to NA] — Cohorts 1-3 and Cohort 4 were conducted as separate studies under the same study protocol. As such, all analyses were conducted separately for Cohorts 1-3 and Cohort 4.
Baseline SCA in Cohort 4 [Median (Inter-Quartile Range); unit: log10 copies/mL] — Baseline HIV-1 RNA levels as detected by single copy assay (SCA) was calculated as the average of the pre-entry and entry SCA measurements for Cohort 4 Population: Cohorts 1-3 were analyzed separately from Cohort 4
  log10 copies/mL
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 3 | 16
    (all) |  |  |  |  | -0.2 [-0.7 to 0.39] | -0.25 [-0.25 to 0.31] | NA [NA to NA] — Cohorts 1-3 and Cohort 4 were conducted as separate studies under the same study protocol. As such, all analyses were conducted separately for Cohorts 1-3 and Cohort 4.
Baseline CA RNA in Cohorts 1-3 [Median (Inter-Quartile Range); unit: log10 copies/mL] — Baseline cell-associated HIV-1 RNA levels (CA-RNA) (log10 copies/mL) were measured in resting CD4 T-cells for Cohorts 1-3. Baseline CA-RNA is the pre-entry measurement for Cohorts 1-3. Population: Cohorts 1-3 were analyzed separately from Cohort 4
  log10 copies/mL
    number analyzed (Participants) | 12 | 12 | 12 | 7 | 0 | 0 | 43
    (all) | 1.9 [1.7 to 2.6] | 2.6 [2.3 to 3] | 2.3 [2.0 to 2.7] | 2.8 [2.4 to 3] |  |  | NA [NA to NA] — Cohorts 1-3 and Cohort 4 were conducted as separate studies under the same study protocol. As such, all analyses were conducted separately for Cohorts 1-3 and Cohort 4.
Baseline CA RNA in Cohort 4 [Median (Inter-Quartile Range); unit: log10 copies/mL] — Baseline cell-associated HIV-1 RNA levels (CA-RNA) (log10 copies/mL) were measured in PBMCs for Cohort 4. Baseline CA-RNA was calculated as the average of the pre-entry and entry CA-RNA measurement for Cohort 4. Population: Cohorts 1-3 were analyzed separately from Cohort 4
  log10 copies/mL
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 3 | 16
    (all) |  |  |  |  | 1.19 [0.9 to 1.64] | 1.61 [1.49 to 2.44] | NA [NA to NA] — Cohorts 1-3 and Cohort 4 were conducted as separate studies under the same study protocol. As such, all analyses were conducted separately for Cohorts 1-3 and Cohort 4.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Grade 3 or Higher Adverse Events (AEs) in Cohorts 1-3 Romidepsin Arms
Description: Proportion of participants with Grade 3 or higher adverse events (AEs) in Cohorts 1-3 Romidepsin Arms, including signs/symptoms, lab toxicities, and /or clinical events probably, possibly, or definitely related to study treatment (as judged by the core team, blinded to treatment arm). The DAIDS AE Grading Table (Version 1.0) was used.
Time Frame: Measured from the time of Romidepsin administration (at entry) until 28 days after the administration
Population: Participants in Cohorts 1-3 who received Romidepsin
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Cohorts 1-3 (Romidepsin): Participants in Cohorts 1-3 received Romidepsin intravenously (IV) over 4 hours (beginning at Hour 0) at the Day 0 study visit.
Arm/Group | Cohorts 1-3 (Romidepsin)
Number analyzed (Participants) | 36
proportion of participants | 0 [0 to 0.097]

2. Primary Outcome: Proportion of Participants With Grade 3 or Higher Adverse Events (AEs) in Cohort 4 Romidepsin Arm
Description: Proportion of participants with Grade 3 or Higher Adverse Events (AEs) in Cohort 4 Romidepsin Arm, including signs/symptoms, lab toxicities, and /or clinical events probably, possibly, or definitely related to study treatment (as judged by the core team, blinded to treatment arm). The DAIDS AE Grading Table (Version 1.0) was used.
Time Frame: Measured from the time of the first Romidepsin administration through 28 days after the last administration (at day 42)
Population: Participants in Cohort 4 who received Romidepsin
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Cohort 4-Arm 4A (Romidepsin): Participants in Cohort 4 received Romidepsin IV over 4 hours (beginning at Hour 0) at the Day 0, 14, 28, and 42 study visits.
Arm/Group | Cohort 4-Arm 4A (Romidepsin)
Number analyzed (Participants) | 13
proportion of participants | 0.077 [0.002 to 0.36]

3. Primary Outcome: Change From Baseline in Plasma HIV-1 RNA Levels as Detected by Single Copy Assay in Cohorts 1-3
Description: Baseline is defined as the average of the pre-entry and entry values. Hour 24/48 is defined as the average of values at 24 and 48 hours after the single administration of Romidepsin or placebo (at study entry).
  Change was calculated as the value at hour 24/48 minus the value at baseline.
Time Frame: Pre-entry, entry, 24 and 48 hours after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Groups:
- Cohorts 1-3 (Romidepsin): Participants in Cohorts 1-3 who received Romidepsin intravenously (IV) over 4 hours (beginning at Hour 0) at the Day 0 study visit.
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
log10 copies/mL | 0.12 [-0.18 to 0.42] | 0.12 [-0.24 to 0.67]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change From Baseline in Plasma HIV-1 RNA Levels as Detected by Single Copy Assay in Cohort 4
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value at 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) minus the value at baseline.
Time Frame: Pre-entry, entry, 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42)
Population: Cohort 4 participants
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
log10 copies/mL
  Change from baseline to 24 hours post infusion 1: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 1 | 0 [-0.32 to 0.23] | -0.11 [-0.45 to 0.55]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | 0.03 [-0.03 to 0.53] | 0.15 [-0.23 to 1.24]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | 0.3 [0 to 0.45] | 0.47 [0.33 to 0.63]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 4 | 0 [-0.17 to 0.23] | 0.33 [0.15 to 0.33]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change From Baseline in Cell-associated HIV-1 RNA Levels in Resting CD4 T-cells in Cohorts 1-3
Description: Baseline is defined as the pre-entry value. Change was calculated as the value at 24 hours after administration of Romidepsin or placebo (at entry) minus the value at baseline.
Time Frame: Pre-entry and 24 hours after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants
Measure: Median (Inter-Quartile Range); unit: log10 (copies/10^6 resting CD4 cells)
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
log10 (copies/10^6 resting CD4 cells) | -.009 [-0.38 to 0.26] | 0 [-0.22 to 0.36]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Change From Baseline in Cell-associated HIV-1 RNA Levels in PBMCs in Cohort 4
Description: as for outcome 4
Time Frame: Pre-entry, entry and 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: log10 (copies/10^6 PBMCs)
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
log10 (copies/10^6 PBMCs)
  Change from baseline to 24 hours post infusion 1 | -0.06 [-0.14 to 0.07] | -0.16 [-0.36 to 0.43]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | -0.07 [-0.38 to 0.31] | -0.52 [-0.91 to -0.15]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | -0.44 [-0.69 to -0.15] | -0.02 [-1.25 to 0.04]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | -0.05 [-0.2 to 0.01] | -0.3 [-0.76 to 0.15]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.92, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA Levels as Detected by Single Copy Assay in Cohorts 1-3
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value at 6 hours, 12 hours, 7 days, 14 days and 28 days after administration of Romidepsin or placebo (at entry) minus the value at baseline.
Time Frame: Pre-entry, entry, 6 hours, 12 hours, 7 days, 14 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
log10 copies/mL
  Change from baseline to 6 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 6 hours post infusion | -0.02 [-0.38 to 0.22] | 0.14 [-0.37 to 0.48]
  Change from baseline to 12 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 12 hours post infusion | 0 [-0.49 to 0.2] | 0.27 [0.14 to 0.57]
  Change from baseline to 7 days post infusion | 0 [-0.25 to 0.39] | 0.27 [-0.16 to 0.63]
  Change from baseline to 14 days post infusion: number analyzed (Participants) | 34 | 7
  Change from baseline to 14 days post infusion | 0 [-0.2 to 0.15] | -0.13 [-0.39 to 0.27]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 28 days post infusion | 0 [-0.3 to 0.3] | -0.08 [-0.3 to 0.09]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 6 hours post infusion; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 12 hours post infusion; Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 14 days post infusion; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA Levels as Detected by Single Copy Assay in Cohort 4
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value at 72 hours after the second administration of Romidepsin or placebo (at day 14) minus the value at baseline.
Time Frame: Pre-entry, entry and 72 hours after the second administration of Romidepsin or placebo (at day 14)
Population: Cohort 4 participants
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 12 | 3
log10 copies/mL | 0 [-0.54 to 0.1] | 0.82 [0.15 to 0.86]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Test type: Superiority; p = 0.029, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in Cell-associated HIV-1 RNA Levels in Resting CD4 T Cells in Cohorts 1-3
Description: Baseline is defined as the pre-entry value. Change was calculated as the value at 14 days after administration of Romidepsin or placebo (at entry) minus the value at baseline.
Time Frame: Pre-entry and 14 days after the administration of RMD or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 34 | 7
log10 copies/mL | 0.02 [-0.42 to 0.31] | -0.05 [-0.38 to 0.46]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Cell-associated HIV-1 RNA Levels in PBMCs in Cohort 4
Description: Baseline is defined as the pre-entry value. Change was calculated as the value at 72 hours after the second administration of Romidepsin or placebo (at day 14) minus the value at baseline.
Time Frame: Pre-entry and 72 hours after the second administration of Romidepsin or placebo (at day 14)
Population: Cohort 4 participants
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 12 | 3
log10 copies/mL | -0.26 [-0.48 to 0.17] | -0.16 [-0.25 to 0.14]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in Histone Acetylation (Median FITC Ac-Histone) in CD3+ Cells in Cohorts 1-3
Description: Baseline is defined as the value at Hour 0, right before the single administration of Romidepsin or placebo.
  Change was calculated as the value at 24 hours after administration of Romidepsin or placebo (at entry) minus the value at baseline.
  Median Fluorescent Intensity (MFI) data describes a shift in the expression of a fluorescently labeled marker on a population of cells. The reported MFI is an arbitrary value dependent on the voltage applied to the corresponding flow cytometer detector.
Time Frame: Hour 0 and 24 hours after the single administration of RMD or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 32 | 6
arbitrary units | -7 [-969 to 1606] | -194 [-1529 to 1343]

12. Secondary Outcome: Change From Baseline in Histone Acetylation in (Median FITC Ac-histone) in CD3+ Cells in Cohort 4
Description: Baseline is defined as the value right before the first administration of Romidepsin or placebo (at entry).
  Change was calculated as the value at 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) and 72 hours after the second administration minus the value at baseline.
  Median Fluorescent Intensity (MFI) data describes a shift in the expression of a fluorescently labeled marker on a population of cells. The reported MFI is an arbitrary value dependent on the voltage applied to the corresponding flow cytometer detector.
Time Frame: Entry, 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42), and 72 hours after the second administration (at day 14)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
arbitrary units
  Change from baseline to 24 hours post infusion 1 | 2402 [1257 to 3821] | 749 [-129 to 1498]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | 2774 [1467 to 5086] | 8497 [696 to 8684]
  Change from baseline to 72 hours post infusion 2: number analyzed (Participants) | 10 | 3
  Change from baseline to 72 hours post infusion 2 | 4741 [3065 to 8518] | 4741 [2479 to 13283]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | 4522 [2388 to 8763] | 5665 [1041 to 7154]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 4 | 4342 [3101 to 26464] | 2697 [937 to 4022]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 72 hours post infusion 2; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change From Baseline in Total HIV-1 DNA in Resting or Total CD4 T Cells in Cohorts 1-3
Description: Baseline is defined as the pre-entry value. Change was calculated as the value at 24 hours and 14 days after administration of Romidepsin or placebo (at entry) minus the value at baseline.
Time Frame: Pre-entry, 24 hours and 14 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: log10 (copies/10^6 resting CD4 cells)
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
log10 (copies/10^6 resting CD4 cells)
  Change from baseline to 24 hours post infusion | -0.04 [-0.18 to 0.06] | 0.05 [-0.41 to 0.19]
  Change from baseline to 14 days post infusion: number analyzed (Participants) | 34 | 7
  Change from baseline to 14 days post infusion | -0.01 [-0.21 to 0.06] | -0.05 [-0.24 to 0.08]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 24 hours post infusion; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 14 days post infusion; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change From Baseline in Total HIV-1 DNA in PBMCs in Cohort 4
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value at 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) and 72 hours after the second administration minus the value at baseline.
Time Frame: Pre-entry, 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) and 72 hours after the second administration (at day 14)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: log10 (copies/10^6 PBMCs)
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
log10 (copies/10^6 PBMCs)
  Change from baseline to 24 hours post infusion 1 | -0.06 [-0.1 to -0.03] | -0.04 [-0.26 to 0.03]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | -0.13 [-0.22 to -0.04] | -0.11 [-0.12 to -0.06]
  Change from baseline to 72 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 72 hours post infusion 2 | -0.13 [-0.25 to -0.05] | -0.07 [-0.25 to -0.04]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | -0.06 [-0.46 to -0.03] | -0.13 [-0.14 to -0.07]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | -0.14 [-0.28 to -0.02] | -0.07 [-0.1 to -0.04]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 72 hours post infusion 2; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: PK Parameters for Romidepsin and Co-administered Antiretroviral Drugs (Efavirenz, Dolutegravir, or Raltegravir) in Cohorts 1-3
Description: Hour 0 is right before the single administration of Romidepsin or placebo (at entry).
  Hour 4 is at the completion of Romidepsin or placebo administration. Hours 6, 12 and 24 are 2, 8 and 20 hours after the completion of Romidepsin or placebo administration.
  PK concentration (ng/mL) for Romidepsin at hours 0, 4, 6, 12 and 24. PK concentration (ng/mL) for co-administered antiretroviral drugs (Efavirenz [EFV], Dolutegravir [DTG], or Raltegravir [RAL]) at hours 0 and 24.
Time Frame: At hours 0, 4, 6, 12 and 24
Population: For Romidepsin PK parameters: Cohorts 1-3 participants who received Romidepsin. For co-administered antiretroviral drugs PK parameters: Cohorts 1-3 participants.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Cohort 1-Arm 1A (Romidepsin) | Cohort 2-Arm 2A (Romidepsin) | Cohort 3-Arm 3A (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 12 | 12 | 12 | 7
ng/mL
  RMD PK concentration at Hour 0: number analyzed (Participants) | 12 | 12 | 12 | 0
  RMD PK concentration at Hour 0 | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) |
  RMD PK concentration at Hour 4: number analyzed (Participants) | 12 | 12 | 12 | 0
  RMD PK concentration at Hour 4 | 12 [6.6 to 16.7] | 75.2 [54.1 to 84] | 89 [53.3 to 127.5] |
  RMD PK concentration at Hour 6: number analyzed (Participants) | 1 | 11 | 12 | 0
  RMD PK concentration at Hour 6 | 3.2 [3.2 to 3.2] | 2.7 [1.7 to 4.2] | 2.6 [2 to 5] |
  RMD PK concentration at Hour 12: number analyzed (Participants) | 12 | 12 | 12 | 0
  RMD PK concentration at Hour 12 | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) |
  RMD PK concentration at Hour 24: number analyzed (Participants) | 12 | 12 | 12 | 0
  RMD PK concentration at Hour 24 | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) | NA [NA to NA] — All 12 participants had concentration <= BQL (below quantifiable limit) |
  EFV PK concentration at Hour 0: number analyzed (Participants) | 8 | 5 | 9 | 3
  EFV PK concentration at Hour 0 | 2030 [1570 to 3750] | 2560 [2490 to 2640] | 2612 [1995 to 3423] | 2520 [2000 to 2758]
  EFV PK concentration at Hour 24: number analyzed (Participants) | 8 | 5 | 9 | 3
  EFV PK concentration at Hour 24 | 2105 [1665 to 3405] | 1870 [1700 to 2390] | 2886 [2262 to 4016] | 1600 [1530 to 1849]
  RAL PK concentration at Hour 0: number analyzed (Participants) | 4 | 5 | 0 | 3
  RAL PK concentration at Hour 0 | 777 [294 to 1990] | 910 [845 to 939] |  | 401 [267 to 726]
  RAL PK concentration at Hour 24: number analyzed (Participants) | 4 | 5 | 0 | 4
  RAL PK concentration at Hour 24 | 1234 [526 to 3475] | 398 [348 to 558] |  | 142 [65 to 390]
  DTG PK concentration at Hour 0: number analyzed (Participants) | 0 | 2 | 3 | 0
  DTG PK concentration at Hour 0 |  | 4035 [2740 to 5330] | 2988 [2163 to 7867] |
  DTG PK concentration at Hour 24: number analyzed (Participants) | 0 | 2 | 2 | 0
  DTG PK concentration at Hour 24 |  | 2190 [1010 to 3370] | 2399 [1181 to 3618] |

16. Secondary Outcome: PK Parameters for Romidepsin and Co-administered Antiretroviral Drugs (Dolutegravir or Raltegravi) in Cohort 4
Description: PK concentration (ng/mL) for Romidepsin pre and post the third and fourth administrations of Romidepsin or placebo.
  PK concentration (ng/mL) for co-administered antiretroviral drugs (Dolutegravir [DTG], or Raltegravir [RAL]) 24 hours after the third and fourth administrations of Romidepsin or placebo.
Time Frame: Pre, post and 24 hours after the third and fourth administrations of Romidepsin or placebo (at days 28 and 42)
Population: For Romidepsin PK parameters: Cohort 4 participants who received the third and fourth Romidepsin infusion.
  For co-administered antiretroviral drugs PK parameters: Cohort 4 participants who received the third and fourth Romidepsin or placebo infusion.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
ng/mL
  RMD PK concentration pre infusion 3: number analyzed (Participants) | 1 | 0
  RMD PK concentration pre infusion 3 | 207 [207 to 207] |
  RMD PK concentration post infusion 3: number analyzed (Participants) | 9 | 0
  RMD PK concentration post infusion 3 | 69 [64 to 164] |
  RMD PK concentration pre infusion 4: number analyzed (Participants) | 11 | 0
  RMD PK concentration pre infusion 4 | NA [NA to NA] — All 11 participants had concentration <= BQL (below quantifiable limit) |
  RMD PK concentration post infusion 4: number analyzed (Participants) | 8 | 0
  RMD PK concentration post infusion 4 | 134 [84 to 211] |
  RAL PK concentration 24 hours post infusion 3: number analyzed (Participants) | 4 | 0
  RAL PK concentration 24 hours post infusion 3 | 906 [119 to 3420] |
  RAL PK concentration 24 hours post infusion 4: number analyzed (Participants) | 4 | 0
  RAL PK concentration 24 hours post infusion 4 | 567 [75 to 2711] |
  DTG PK concentration 24 hours post infusion 3: number analyzed (Participants) | 7 | 3
  DTG PK concentration 24 hours post infusion 3 | 2124 [1147 to 3865] | 913 [274 to 1128]
  DTG PK concentration 24 hours post infusion 4: number analyzed (Participants) | 7 | 3
  DTG PK concentration 24 hours post infusion 4 | 1568 [985 to 2779] | 833 [274 to 1323]

17. Secondary Outcome: HIV-1 RNA Levels in Cohorts 1-3
Description: HIV-1 RNA levels at 7 days after the single administration of Romidepsin or placebo (at entry)
Time Frame: 7 days after the administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Arm 1A (Romidepsin) | Cohort 2-Arm 2A (Romidepsin) | Cohort 3-Arm 3A (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 12 | 12 | 12 | 7
Participants
  < 40 copies/mL | 11 | 12 | 12 | 7
  40-199 copies/mL | 1 | 0 | 0 | 0

18. Secondary Outcome: HIV-1 RNA Levels in Cohort 4
Description: HIV-1 RNA levels at 7 days after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42)
Time Frame: 7 days after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42)
Population: Cohort 4 participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
Participants
  HIV-1 RNA level at day 7 post infusion 1: number analyzed (Participants) | 13 | 2
  HIV-1 RNA level at day 7 post infusion 1: < 40 copies/mL | 13 | 2
  HIV-1 RNA level at day 7 post infusion 1: 40 - 199 copies/mL | 0 | 0
  HIV-1 RNA level at day 7 post infusion 2: number analyzed (Participants) | 8 | 3
  HIV-1 RNA level at day 7 post infusion 2: < 40 copies/mL | 8 | 3
  HIV-1 RNA level at day 7 post infusion 2: 40 - 199 copies/mL | 0 | 0
  HIV-1 RNA level at day 7 post infusion 3: number analyzed (Participants) | 11 | 3
  HIV-1 RNA level at day 7 post infusion 3: < 40 copies/mL | 11 | 3
  HIV-1 RNA level at day 7 post infusion 3: 40 - 199 copies/mL | 0 | 0
  HIV-1 RNA level at day 7 post infusion 4: number analyzed (Participants) | 11 | 3
  HIV-1 RNA level at day 7 post infusion 4: < 40 copies/mL | 11 | 3
  HIV-1 RNA level at day 7 post infusion 4: 40 - 199 copies/mL | 0 | 0

19. Secondary Outcome: Number of Participants With Reported Grade 2-4 AEs in Cohorts 1-3
Description: Number of participants with reported grade 2-4 adverse events including signs/symptoms, lab toxicities, and clinical events that are at least possibly related to study treatment. The DAIDS AE Grading Table (Version 1.0) was used.
Time Frame: Measured from study entry to off study
Population: Cohorts 1-3 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Arm 1A (Romidepsin) | Cohort 2-Arm 2A (Romidepsin) | Cohort 3-Arm 3A (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 12 | 12 | 12 | 7
Participants | 4 | 2 | 1 | 1

20. Secondary Outcome: Number of Participants With Reported Grade 2-4 AEs in Cohort 4
Description: as for outcome 19
Time Frame: Measured from study entry to off study
Population: Cohort 4 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
Participants | 5 | 0

21. Secondary Outcome: Change From Baseline in CD4+ and CD8+ T Cell Percent in Cohorts 1-3
Description: Change in CD4+ and CD8+T cell percent from baseline to after the single administration of Romidepsin or placebo
Time Frame: Measured through participant's last study visit
Population: Cohorts 1-3 participants did not have CD4+ and CD8+ T cell percent collected
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in CD4+ T Cell Percent in Cohort 4
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value at 24 hours post each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) and 2, 5, 10 and 18 weeks post the fourth administration minus the value at baseline
Time Frame: Pre-entry, entry, 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42), and 2, 5, 10 and 18 weeks after the fourth administration (at day 42)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD4 cells
  Change from baseline to 24 hours post infusion 1 | -2.5 [-3.5 to -0.5] | -2 [-2 to 2.5]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | -4.5 [-5.9 to -2.4] | 0.5 [-1 to 2]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | -3.5 [-6.5 to -2.5] | 1 [-0.5 to 3]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 4 | -4.5 [-7.5 to -2.5] | 0.5 [0 to 3]
  Change from baseline to 2 weeks post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 2 weeks post infusion 4 | -0.5 [-4.8 to 0.5] | -0.5 [-1 to 2]
  Change from baseline to 5 weeks post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 5 weeks post infusion 4 | -1.8 [-3 to -0.4] | 0 [-2.5 to 0]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 10 weeks post infusion 4 | -2.8 [-3.5 to -1.5] | -0.5 [-4 to 2]
  Change from baseline to 18 weeks post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 18 weeks post infusion 4 | -0.5 [-3.2 to 1.1] | -2.5 [-6 to 1]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 2 weeks post infusion 4; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 5 weeks post infusion 4; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 18 weeks post infusion 4; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Change From Baseline in CD8+ T Cell Percent in Cohort 4
Description: Change in CD8+ T cell percent from baseline to after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42)
Time Frame: Measured through 28 days after the single administration of RMD or placebo (at entry, and days 14, 28 and 42)
Population: Cohort 4 participants did not have CD8+ T cell percent collected
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD38/HLA-DR Expression on CD4+ T-cells) in Cohorts 1-3
Description: Baseline is defined as the value at hour 0, where hour 0 is right before the single administration of Romidepsin or placebo (at entry).
  Change was calculated as the value at 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo minus the value at baseline.
Time Frame: Hour 0 and 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD4 cells
  Change from baseline to 48 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 48 hours post infusion | 0.5 [-0.3 to 1.8] | 0.4 [-1.2 to 2.8]
  Change from baseline to 7 days post infusion | 1 [-0.1 to 2.7] | -1 [-2 to 0.8]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 34 | 7
  Change from baseline to 28 days post infusion | 1.2 [-3.2 to 2.6] | -1.4 [-2.4 to 0.2]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 48 hours post infusion; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD38/HLA-DR Expression on CD8+ T-cells) in Cohorts 1-3
Description: as for outcome 24
Time Frame: Hour 0 and 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD8 cells
  Change from baseline to 48 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 48 hours post infusion | 0.1 [-1.2 to 1.8] | 0.3 [-0.9 to 1.3]
  Change from baseline to 7 days post infusion | 0.8 [-0.8 to 3] | -1.3 [-2 to -0.4]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 34 | 7
  Change from baseline to 28 days post infusion | 0.3 [-4.2 to 3.1] | -0.1 [-2.7 to 2.4]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 48 hours post infusion; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD69/CD25 Expression on CD4+ T-cells) in Cohorts 1-3
Description: as for outcome 24
Time Frame: Hour 0 and 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD4 cells
  Change from baseline to 48 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 48 hours post infusion | 0 [-0.1 to 0.2] | 0 [-0.1 to 0.2]
  Change from baseline to 7 days post infusion | 0 [-0.1 to 0.3] | 0 [-0.1 to 0.4]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 34 | 7
  Change from baseline to 28 days post infusion | 0 [-0.1 to 0.1] | 0 [0 to 0.4]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 48 hours post infusion; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD69/CD25 Expression on CD8+ T-cells) in Cohorts 1-3
Description: as for outcome 24
Time Frame: Hour 0 and 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD8 cells
  Change from baseline to 48 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 48 hours post infusion | 0 [0 to 0.1] | 0 [-0.1 to 0.1]
  Change from baseline to 7 days post infusion | 0 [-0.1 to 0.1] | 0 [-0.1 to 0.1]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 34 | 7
  Change from baseline to 28 days post infusion | 0 [-0.1 to 0.1] | 0 [-0.1 to 0]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 48 hours post infusion; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.92, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD38/HLA-DR Expression on CD4+ T-cells) in Cohort 4
Description: Baseline is defined as the average of the two pre-entry values. Change was calculated as the value at 24 hours post first and fourth administration of Romidepsin or placebo (at entry and day 42) and 10 weeks post the fourth administration (at day 42) minus the value at baseline.
Time Frame: Pre-entry, 24 hours after the first and fourth administration of Romidepsin or placebo (at entry and day 42), and 10 weeks after the fourth administration (at day 42)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD4 cells
  Change from baseline to 24 hours post infusion 1: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 1 | 0.2 [-0.1 to 1.2] | 0.5 [-1.4 to 1.1]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | 1 [0.4 to 3.5] | 2 [1.6 to 2.3]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 10 | 3
  Change from baseline to 10 weeks post infusion 4 | 0.4 [-0.5 to 1.3] | 0.7 [0.6 to 2.2]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD38/HLA-DR Expression on CD8+ T-cells) in Cohort 4
Description: as for outcome 28
Time Frame: as for outcome 28
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD8 cells
  Change from baseline to 24 hours post infusion 1: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 1 | 0.6 [-0.2 to 1.8] | 0.2 [-0.2 to 0.2]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | 1.1 [-0.5 to 2.1] | 1.1 [-0.3 to 2.4]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 10 | 3
  Change from baseline to 10 weeks post infusion 4 | -0.3 [-2.8 to 0.4] | 2.8 [1.6 to 8.7]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); hange from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD69/CD25 Expression on CD4+ T-cells) in Cohort 4
Description: Baseline is defined as the average of the two pre-entry values. Change was calculated as the value at 24 hours post first and fourth administration of Romidepsin or placebo (at etnry and day 42) and 10 weeks post the fourth administration (at day 42) minus the value at baseline.
Time Frame: Pre-entry, 24 hours after the first and fourth administration of Romidepsin or placebo (at etnry and day 42), and 10 weeks after the fourth administration (at day 42)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD4 cells
  Change from baseline to 24 hours post infusion 1: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 1 | 0 [0 to 0.1] | -0.1 [-0.1 to 0.1]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | 0 [0 to 0.4] | -0.1 [-0.1 to 0]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 10 | 3
  Change from baseline to 10 weeks post infusion 4 | 0 [-0.2 to 0.5] | -0.1 [-0.1 to 0.1]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Change From Baseline in Cellular Markers of Immune Activation (CD69/CD25 Expression on CD8+ T-cells) in Cohort 4
Description: as for outcome 30
Time Frame: Pre-entry, 24 hours after the first and fourth administration of Romidepsin or placebo (at etnry and day 42), and 10 weeks after the fourth administration (at day 42
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD8 cells
  Change from baseline to 24 hours post infusion 1: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 1 | 0 [0 to 0.1] | 0 [-0.1 to 0]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | 0 [0 to 0.1] | -0.1 [-0.2 to 0]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 10 | 3
  Change from baseline to 10 weeks post infusion 4 | 0 [0 to 0.1] | 0 [-0.2 to 0]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Change From Baseline in Percentage of CD4+ T-cells Expressing Annexin V and/or 7 Amino-actinomycin D (7-AAD) in Cohorts 1-3
Description: Baseline is defined as the value at hour 0, where hour 0 is right before the single administration of Romidepsin or placebo (at entry).
  Change was calculated as the value at 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry) minus the value at baseline.
Time Frame: Hour 0 and 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD4 cells
  Change from baseline to 48 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 48 hours post infusion | 0.2 [-0.6 to 1] | 1.2 [0.1 to 7]
  Change from baseline to 7 days post infusion | 0.6 [-1.2 to 2] | 0 [-3.7 to 0.3]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 28 days post infusion | 1.2 [0.1 to 3.9] | -1.3 [-3.6 to 0.1]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 48 hours post infusion; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Change From Baseline in Percentage of CD8+ T-cells Expressing Annexin V and/or 7 Amino-actinomycin D (7-AAD) in Cohorts 1-3
Description: as for outcome 32
Time Frame: Hour 0 and 48 hours, 7 days and 28 days after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD8 cells
  Change from baseline to 48 hours post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 48 hours post infusion | -0.1 [-2.1 to 0.6] | 1.8 [-1 to 4.3]
  Change from baseline to 7 days post infusion | 0.3 [-1.4 to 3.1] | -1.1 [-4.6 to 3.3]
  Change from baseline to 28 days post infusion: number analyzed (Participants) | 35 | 7
  Change from baseline to 28 days post infusion | 0.9 [-1.7 to 3] | -1.9 [-4.1 to 2.5]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 48 hours post infusion; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 7 days post infusion; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change from baseline to 28 days post infusion; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Change From Baseline in Percentage of CD4+ T-cells Expressing Annexin V and/or 7 Amino-actinomycin D (7-AAD) in Cohort 4
Description: as for outcome 28
Time Frame: as for outcome 28
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD4 cells
  Change from baseline to 24 hours post infusion 1 | 0.5 [-2.7 to 1.3] | -1.4 [-2.2 to 7]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 4 | -2 [-4.5 to 3.1] | 0.9 [-0.7 to 2.4]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 10 | 3
  Change from baseline to 10 weeks post infusion 4 | 0.3 [-2.9 to 1.5] | 0.1 [-3.7 to 5.8]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Change From Baseline in Percentage of CD8+ T-cells Expressing Annexin V and/or 7 Amino-actinomycin D (7-AAD) in Cohort 4
Description: as for outcome 28
Time Frame: as for outcome 28
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD8 cells
  Change from baseline to 24 hours post infusion 1 | 0.1 [-3.7 to 1.3] | -4.1 [-5.1 to 8]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 4 | -2.5 [-3.3 to 15.4] | -.6 [-1.5 to 0.3]
  Change from baseline to 10 weeks post infusion 4: number analyzed (Participants) | 10 | 3
  Change from baseline to 10 weeks post infusion 4 | 0.9 [-4.1 to 4.3] | -0.8 [-6.5 to 10.2]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 10 weeks post infusion 4; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Change From Baseline in PTEF-b Phosphorylation (pNFKB+% and pS175%) in CD4+ T-cells in Cohorts 1-3
Description: Baseline is defined as the value at hour 0, where hour 0 is right before the single administration of Romidepsin or placebo (at entry).
  Change was calculated as the value at 24 hours after the single administration of Romidepsin or placebo (at entry) minus the value at baseline.
Time Frame: Hour 0 and 24 hours after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD4 cells
  Change in pNFKB+% on CD4: number analyzed (Participants) | 35 | 7
  Change in pNFKB+% on CD4 | 20 [9.4 to 35.1] | 19.3 [2.4 to 39.1]
  Change in pS175% on CD4: number analyzed (Participants) | 35 | 7
  Change in pS175% on CD4 | 18.1 [8.5 to 28.3] | 6 [-3.5 to 31.5]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change in pNFKB+% on CD4; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change in pS175% on CD4; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Change From Baseline in PTEF-b Phosphorylation (pNFKB+% and pS175%) in CD8+ T-cells in Cohorts 1-3
Description: as for outcome 36
Time Frame: Hour 0 and 24 hours after the single administration of Romidepsin or placebo (at entry)
Population: Cohorts 1-3 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD8 cells
Arm/Group | Cohorts 1-3 (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin)
Number analyzed (Participants) | 36 | 7
percentage of CD8 cells
  Change in pNFKB+% on CD8: number analyzed (Participants) | 35 | 7
  Change in pNFKB+% on CD8 | 16.5 [1.4 to 29] | 3.8 [-8.3 to 29.9]
  Change in pS175% on CD8: number analyzed (Participants) | 35 | 7
  Change in pS175% on CD8 | 26.5 [18.1 to 38.8] | 25.3 [14.9 to 37.2]
Statistical Analysis 1: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change in pNFKB+% on CD8; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohorts 1-3 (Romidepsin) vs Cohorts 1-3 (Placebo for Romidepsin); Change in pS175% on CD8; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

38. Secondary Outcome: Change From Baseline in PTEF-b Phosphorylation (pNFKB+%) in CD4+ T-cells in Cohort 4
Description: Baseline is defined as the average of the pre-entry and entry values. Change was calculated as the value at 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) and 72 hours after the second administration (at day 14) minus the value at baseline.
Time Frame: Pre-entry, entry, 24 hours after each administration of Romidepsin or placebo (at entry, and days 14, 28 and 42) and 72 hours after the second administration (at day 14)
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD4 cells
  Change from baseline to 24 hours post infusion 1 | 5.04 [0 to 8.63] | 0.01 [0 to 0.01]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | 8.78 [4.77 to 13.69] | 0 [0 to 0.03]
  Change from baseline to 72 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 72 hours post infusion 2 | 6.39 [0 to 9.83] | 0 [0 to 0.02]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | 5.78 [0.02 to 11.22] | 0 [0 to 0.08]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | 9.63 [4.95 to 11.74] | 0 [-0.01 to 0]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 72 hours post infusion 2; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Change From Baseline in PTEF-b Phosphorylation (pS175+%) in CD4+ T-cells in Cohort 4
Description: as for outcome 38
Time Frame: as for outcome 38
Population: Cohort 4 participants with available data
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
Number analyzed (Participants) | 13 | 3
percentage of CD4 cells
  Change from baseline to 24 hours post infusion 1 | 9.93 [0.01 to 17.06] | -0.01 [-0.01 to 0.01]
  Change from baseline to 24 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 24 hours post infusion 2 | 17 [12.87 to 18.66] | -0.01 [-0.01 to 0]
  Change from baseline to 72 hours post infusion 2: number analyzed (Participants) | 12 | 3
  Change from baseline to 72 hours post infusion 2 | 11 [0.01 to 15.36] | -0.01 [-0.01 to 0]
  Change from baseline to 24 hours post infusion 3: number analyzed (Participants) | 11 | 3
  Change from baseline to 24 hours post infusion 3 | 14.85 [5.29 to 15.58] | 0 [-0.01 to 0.05]
  Change from baseline to 24 hours post infusion 4: number analyzed (Participants) | 11 | 2
  Change from baseline to 24 hours post infusion 4 | 16.52 [6.82 to 18.21] | 0.01 [0 to 0.02]
Statistical Analysis 1: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 1; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 2; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 72 hours post infusion 2; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 3; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cohort 4-Arm 4A (Romidepsin) vs Cohort 4-Arm 4B (Placebo for Romidepsin); Change from baseline to 24 hours post infusion 4; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from study entry until the end of study (28 days for Cohorts 1-3 and up to 48 weeks for Cohort 4).
Description: The protocol required reporting of all diagnoses, all signs/symptoms/laboratory values Grade ≥ 2, and all signs/symptoms/laboratory values that led to treatment change and/or Grade ≥ 3 and/or met EAE or ICH reporting requirements. For grading, sites referred to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009), http://rsc.tech-res.com/clinical-research-sites/safety-reporting.
Arm/Group | Cohort 1-Arm 1A (Romidepsin) | Cohort 2-Arm 2A (Romidepsin) | Cohort 3-Arm 3A (Romidepsin) | Cohorts 1-3 (Placebo for Romidepsin) | Cohort 4-Arm 4A (Romidepsin) | Cohort 4-Arm 4B (Placebo for Romidepsin)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/7 | 0/13 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/7 | 0/13 | 1/3
Other Adverse Events (participants affected / at risk) | 8/12 | 6/12 | 1/12 | 3/7 | 9/13 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1-Arm 1A (Romidepsin) (N=12) | Cohort 2-Arm 2A (Romidepsin) (N=12) | Cohort 3-Arm 3A (Romidepsin) (N=12) | Cohorts 1-3 (Placebo for Romidepsin) (N=7) | Cohort 4-Arm 4A (Romidepsin) (N=13) | Cohort 4-Arm 4B (Placebo for Romidepsin) (N=3)
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1-Arm 1A (Romidepsin) (N=12) | Cohort 2-Arm 2A (Romidepsin) (N=12) | Cohort 3-Arm 3A (Romidepsin) (N=12) | Cohorts 1-3 (Placebo for Romidepsin) (N=7) | Cohort 4-Arm 4A (Romidepsin) (N=13) | Cohort 4-Arm 4B (Placebo for Romidepsin) (N=3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Abscess bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 1 | 0 | 3 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT interval normal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Haemoglobin abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint noise (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 3 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT01933594/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT01933594/SAP_000.pdf